CLINICAL TRIAL: NCT03630354
Title: EXERCISING TOGETHER © for Couples Coping With Cancer
Brief Title: EXERCISING TOGETHER for Couples Coping With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00018000; NCI-2018-01404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018000 (Other: OHSU Knight Cancer Institute); R01CA218093 (NIH)
Record Dates: First submitted 2018-08-03; First posted 2018-08-14 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Carcinoma; Colorectal Carcinoma; Malignant Solid Neoplasm; Prostate Carcinoma; Stage I Colorectal Cancer AJCC v8; Stage I Prostate Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (supervised exercise together) (Experimental): Couples perform partnered exercise over 1 hour, 2 days per week in a supervised, group setting remotely for 6 months.
  Interventions: Behavioral: Exercise Intervention (supervised); Other: Questionnaire Administration
- Arm II (supervised exercise separately) (Experimental): Survivors and partners perform exercise routines over 1 hour, 2 days per week separately in a supervised group setting remotely for 6 months.
  Interventions: Behavioral: Exercise Intervention (supervised); Other: Questionnaire Administration
- Arm III (unsupervised exercise separately) (Experimental): Survivors and partners undergo 2 training sessions remotely over 1 hour with an exercise trainer and then perform exercise routines over 1 hour, 2 days per week unsupervised at home or a facility following an instructional DVD.
  Interventions: Behavioral: Exercise Intervention (unsupervised); Other: Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention (supervised) — Complete supervised exercise
  Arms: Arm I (supervised exercise together); Arm II (supervised exercise separately)
Behavioral: Exercise Intervention (unsupervised) — Complete unsupervised exercise
  Arms: Arm III (unsupervised exercise separately)
Other: Informational Intervention — Receive instructional DVD
  Arms: Arm III (unsupervised exercise separately)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The Exercising Together trial is a single-blind, parallel group, randomized controlled trial comparing 3 arms: Arm 1 (experimental): Exercising Together where couples perform partnered exercise in a supervised, group setting versus two comparator conditions where survivors and partners perform exercise routines separately in either a supervised group setting (Arm 2) or unsupervised at home (Arm 3). All three arms will train for a 6-month period and then be followed 6 months later. Data will be collected at baseline, 3, 6 and 12 months.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of Exercising Together on relationship quality (intimacy, communication and incongruence) in couples coping with prostate cancer (PC), breast cancer (BC), or colorectal cancer (CRC).

II. Determine the efficacy of Exercising Together on the physical health (body composition, lipids, insulin resistance, blood pressure, inflammation, and physical function) and mental health (anxiety, depressive symptoms, fear of recurrence) of both the survivor and spouse/partner.

III. Determine how long individual and couple-level benefits from Exercising Together last.

EXPLORATORY OBJECTIVE:

I. Identify the types of couples that benefit most from Exercising Together.

OUTLINE: Study is a 3-group, 12-month (6 months of exercise training + 6-months follow-up) randomized trial.

ARM I: Exercising Together Program: Couples perform partnered exercise over 1 hour, 2 days per week in a supervised, group setting.

ARM II: Exercising Together Program: Survivors and spouses/partners perform exercise routines separately in a supervised group setting

ARM III: Survivors and partners undergo 2 training sessions over 1 hour with an exercise trainer and then perform exercise routines over 1 hour 2 days per week separately unsupervised at home or a facility following an instructional digital video disc (DVD).

The basic training program for all three study arms is a functional strength training program. Participants will use free weights (weighted vest, dumbbells, elastic bands) while performing lower body (chair rises, squats, lunges, stepups) and upper body (1-arm row, bench press, push-ups, triceps extension, bicep curls, shoulder raise) resistance exercise. Volume of resistance exercise, determined by intensity (weight, tailored to each individual) and duration (number of repetitions and sets), is gradually increased from low weight and high repetitions to more weight and fewer repetitions over the training period.

ELIGIBILITY:
Inclusion Criteria:

* SURVIVORS ONLY:
* Histologically confirmed PC, BC or CRC without evidence of metastatic disease (confirmed by self-report on Health History Questionnaire. In the case a participant isn't able to confirm this criterion, a letter will be sent to his or her physician)
* Three years or less from diagnosis date, by month and year, at time of enrollment (confirmed by self-report on Health History Questionnaire. In the case a participant isn't able to confirm this criterion, a letter will be sent to his or her physician)
* Completed treatment (e.g., surgery, radiation and/or chemotherapy) >= 6 weeks prior to enrollment. Concurrent adjuvant hormone therapy is permitted and must have been initiated >= 6 weeks prior to enrollment. For prostate cancer, androgen deprivation therapy (ADT) may constitute primary treatment and must have been initiated >= 6 weeks prior to enrollment. For breast cancer, hormone therapy may constitute primary treatment and must have been initiated >= 6 weeks prior to enrollment. (confirmed by self-report on Health History Questionnaire. In the case a participant isn't able to confirm this criterion, a letter will be sent to his or her physician)
* Co-residing with an intimate partner or spouse who is willing to participate (confirmed by self-report on Health History Questionnaire)
* SURVIVORS AND SPOUSES/PARTNERS:
* Underactive (< 2 strength training sessions per week, lasting 30 minutes or more per session, at a moderate intensity in the last month) (confirmed by self-report on Health History Questionnaire or by discretion of the principal investigator)

Exclusion Criteria:

* SURVIVORS AND SPOUSES/PARTNERS
* Cognitive difficulties that preclude answering the survey questions, participating in the exercise classes or performance tests, or providing informed consent as determined by the professional opinion of the principal investigator, Dr. Kerri Winters-Stone
* A medical condition, movement or neurological disorder, or medication use that contraindicates participation in moderate intensity exercise. Specific contraindications include the following: declared pregnancy, poorly controlled diabetes, recent cardiac event, neuromuscular disease, untreated orthostatic hypertension, recent surgery, acute hernia, acute rheumatoid arthritis, severe memory disorders, severe balance disorder, inability to ambulate (use of an assistive device permitted), inability to stand for 3 minutes, severe hearing or vision problem. (For Survivor: Confirmed by physician clearance; For Spouse/Partner: must answer 'No' to American College of Sports Medicine pre-participation screening questions. If spouse/partner answers 'Yes' to either question they will be considered eligible upon physician clearance. Physician clearance may also be requested at the discretion of the principal investigator. For either: absence of pregnancy in persons who could possibly be pregnant but have not declared a pregnancy at screening, will be further screened with a pregnancy test administered at each testing visit.)
* Knowingly unable to attend > 75% of the intervention classes due to conflict with the designated time of day, days of the week, and/or location for the exercise class which they initially enrolled. (Confirmed by documentation in the Case Report Form titled "CRF - Participant Contact Info_Exercising Together")
* Not fluent in English and therefore incapable of answering survey questions, participating in class, following directions during performance testing, and providing informed consent when English is the language used. (Confirmed by documentation in the Case Report Form titled "CRF - Participant Contact Info_Exercising Together" or the professional opinion of the Principal Investigator, Dr. Kerri Winters-Stone.)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual quantitative participant data collected during the trial, after deidentification.
Time Frame: Beginning 3 months following final publication.
Access Criteria: Access will be provided to investigators who provide a methodologically sound proposal and complete a data sharing agreement that includes commitments to: (1) using the data only for research purposes and not to identify any individual participant, (2) securing the data using appropriate computer technology, and (3) destroying or returning the data after analyses are completed.
  Proposals should be directed to wintersk@ohsu.edu. To gain access to data, data requestors will need to sign a data sharing agreement.

REFERENCES:
- [Derived] Skiba MB, Dieckmann NF, Lyons KS, Winters-Stone KM. Associations between perceptions of relationship quality and markers of inflammation and insulin resistance among couples coping with cancer. J Cancer Surviv. 2023 Aug;17(4):957-966. doi: 10.1007/s11764-022-01299-5. Epub 2022 Nov 26. PMID 36435952
- [Derived] Winters-Stone KM, Boisvert C, Li F, Lyons KS, Beer TM, Mitri Z, Meyers G, Eckstrom E, Campbell KL. Delivering exercise medicine to cancer survivors: has COVID-19 shifted the landscape for how and who can be reached with supervised group exercise? Support Care Cancer. 2022 Mar;30(3):1903-1906. doi: 10.1007/s00520-021-06669-w. Epub 2021 Nov 6. PMID 34741653
- [Derived] Winters-Stone KM, Lyons KS, Dieckmann NF, Lee CS, Mitri Z, Beer TM. Study protocol for the Exercising Together(c) trial: a randomized, controlled trial of partnered exercise for couples coping with cancer. Trials. 2021 Aug 30;22(1):579. doi: 10.1186/s13063-021-05548-3. PMID 34461975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Community-dwelling couples were recruited between January 2019 and October 2022. The first couple was enrolled on January 18, 2019 and the last was couple was enrolled on October 26, 2022.
Pre-assignment Details: Of 269 consented couples, 248 couples (496 individuals: 248 survivors + 248 partners) met inclusion criteria and were randomized to an intervention group.
Groups:
- Arm I (Supervised Exercise Together): Couples perform partnered exercise over 1 hour, 2 days per week in a supervised, group setting remotely for 6 months.
  Exercise Intervention: Complete supervised exercise
  Questionnaire Administration: Ancillary studies
- Arm II (Supervised Exercise Separately): Survivors and partners perform exercise routines over 1 hour, 2 days per week separately in a supervised group setting remotely for 6 months.
  Exercise Intervention: Complete supervised exercise
  Questionnaire Administration: Ancillary studies
- Arm III (Unsupervised Exercise Separately): Survivors and partners undergo 2 training sessions remotely over 1 hour with an exercise trainer and then perform exercise routines over 1 hour, 2 days per week unsupervised at home or a facility following an instructional DVD.
  Exercise Intervention: Complete unsupervised exercise
  Informational Intervention: Receive instructional DVD
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Started | 164 (82 survivors and 82 partners) | 170 (85 survivors and 85 partners) | 162 (81 survivors and 81 partners)
Completed | 148 (74 survivors and 74 partners) | 148 (74 survivors and 74 partners) | 126 (63 survivors and 63 partners)
Not Completed | 16 | 22 | 36

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants reflect total number of individuals (survivors + partners).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately) | Total
Number analyzed (Participants) | 164 | 170 | 162 | 496
Age, Continuous [Mean (Standard Deviation); unit: years] — Survivors Population: Survivors only
  years
    number analyzed (Participants) | 82 | 85 | 81 | 248
    (all) | 64.6 (9.53) | 62.6 (10.9) | 62.9 (10.5) | 63.3 (10.4)
Age, Continuous [Mean (Standard Deviation); unit: years] — Partners Population: Partners only
  years
    number analyzed (Participants) | 82 | 85 | 81 | 248
    (all) | 64.8 (9.46) | 62.7 (10.7) | 62.6 (65.5) | 63.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Survivors Population: Survivors only
  Participants
    number analyzed (Participants) | 82 | 85 | 81 | 248
    Female | 42 | 45 | 46 | 133
    Male | 40 | 40 | 35 | 115
Sex: Female, Male [Count of Participants; unit: Participants] — Partners Population: Partners only
  Participants
    number analyzed (Participants) | 82 | 85 | 81 | 248
    Female | 41 | 43 | 39 | 123
    Male | 41 | 42 | 42 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Survivors Population: Survivors only
  Participants
    number analyzed (Participants) | 82 | 85 | 81 | 248
    Hispanic or Latino | 3 | 1 | 3 | 7
    Not Hispanic or Latino | 78 | 82 | 78 | 238
    Unknown or Not Reported | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Partners Population: Partners only
  Participants
    number analyzed (Participants) | 82 | 85 | 81 | 248
    Hispanic or Latino | 3 | 1 | 4 | 8
    Not Hispanic or Latino | 79 | 84 | 75 | 238
    Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Survivors Population: Survivors only
  Participants
    number analyzed (Participants) | 82 | 85 | 81 | 248
    American Indian or Alaska Native | 0 | 1 | 0 | 1
    Asian | 0 | 3 | 5 | 8
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
    Black or African American | 1 | 0 | 1 | 2
    White | 77 | 75 | 72 | 224
    More than one race | 3 | 4 | 2 | 9
    Unknown or Not Reported | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Partners Population: Partners only
  Participants
    number analyzed (Participants) | 82 | 85 | 81 | 248
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 2 | 3 | 4 | 9
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
    Black or African American | 2 | 0 | 1 | 3
    White | 75 | 78 | 70 | 223
    More than one race | 2 | 2 | 3 | 7
    Unknown or Not Reported | 0 | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants] — Survivors Population: Survivors only
  Participants
    United States: number analyzed (Participants) | 82 | 85 | 81 | 248
    United States | 82 | 85 | 81 | 248
Region of Enrollment [Count of Participants; unit: Participants] — Partners Population: Partners only
  Participants
    United States: number analyzed (Participants) | 82 | 85 | 81 | 248
    United States | 82 | 85 | 81 | 248

OUTCOME MEASURES:

1. Primary Outcome: Dyadic Coping - Active Engagement
Description: Measured by the Active Engagement subscale from the Relationship Focused Coping Scale. The subscale assesses the degree with which couples practice active engagement by responding to five items on a Likert scale from 1 (never) to 5 (very often). Scores range from 5 to 25, with higher scores indicating more active engagement. Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -0.45 [-1.16 to 0.27] | 0.81 [0.11 to 1.50] | 0.07 [-0.68 to 0.83]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.35 [-1.01 to 0.30] | -0.61 [-1.26 to 0.03] | -0.08 [-0.79 to 0.63]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | 0.05 [-0.61 to 0.71] | -0.08 [-0.72 to 0.57] | -0.91 [-1.62 to -0.19]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -0.52 [-1.20 to 0.16] | -0.14 [-0.81 to 0.54] | -0.35 [-1.09 to 0.39]

2. Primary Outcome: Dyadic Coping - Protective Buffering
Description: Measured by the Protective Buffering Subscale from the Relationship Focused Coping Scale. Assesses the degree with which couples practice protective buffering by responding to six items using a Likert scale of 1 (never) to 5 (very often). Scores range from 6 to 30 with higher scores indicating more protective buffering. Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6, and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -0.48 [-1.24 to 0.29] | -0.18 [-0.93 to 0.57] | -0.13 [-0.93 to 0.66]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.21 [-0.91 to 0.50] | -0.46 [-1.16 to 0.24] | -0.57 [-1.34 to 0.20]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | 0.36 [-0.39 to 1.10] | -0.09 [-0.81 to 0.62] | 0.36 [-0.44 to 1.15]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -0.04 [-0.75 to 0.68] | -0.20 [-0.91 to 0.51] | -0.27 [-1.07 to 0.54]

3. Primary Outcome: Emotional Intimacy
Description: Measured by the 7-item Dyadic Adjustment Scale (DAS) to assess each partner's satisfaction with their relationship by answering 7 questions on a 6-point scale ranging from 1(always agree) to 6 (always disagree). Scores range from 0-21 with higher scores indicating better dyadic adjustment. Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | 3.37 [.78 to 5.97] | 2.61 [.06 to 5.15] | 2.97 [.20 to 5.73]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -2.87 [-5.84 to .10] | -2.30 [-5.26 to .67] | -1.33 [-4.66 to 2.01]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | .98 [-1.25 to 3.20] | 1.90 [-.24 to 4.05] | -.99 [-3.42 to 1.43]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -2.63 [-5.01 to -.26] | -.43 [-2.73 to 1.88] | 1.96 [-.64 to 4.56]

4. Primary Outcome: Physical Intimacy - Engagement in Sex
Description: Measured by the Physical Intimacy Behavior scale which asks participants the frequency that they engage in sexual behaviors answering two questions on a scale from 1 (none of the time) to 4 (most or all of the time). Scores range from 2 to 8 with higher scores indicating higher physical intimacy.
Time Frame: Baseline, 3, 6 and 12 months
Population: This measure had a significant amount of missing data (due to the sensitivity of the questions) so the total sample size is reduced.
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 151 | 161 | 138
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 73 | 81 | 69
  Survivor: Baseline-6mo | 0.08 [-0.23 to 0.40] | -0.04 [-0.34 to 0.26] | -0.07 [-0.42 to 0.29]
  Survivor: 6mo-12mo: number analyzed (Participants) | 73 | 81 | 69
  Survivor: 6mo-12mo | -0.02 [-0.29 to 0.24] | 0.19 [-0.07 to 0.44] | -0.02 [-0.32 to 0.28]
  Partner: Baseline-6mo: number analyzed (Participants) | 78 | 80 | 69
  Partner: Baseline-6mo | 0.10 [-0.20 to 0.39] | 0.16 [-0.11 to 0.43] | -0.08 [-0.41 to 0.24]
  Partner: 6mo-12mo: number analyzed (Participants) | 78 | 80 | 69
  Partner: 6mo-12mo | -0.12 [-0.41 to 0.17] | -0.23 [-0.50 to 0.05] | 0.03 [-0.30 to 0.35]

5. Primary Outcome: Physical Intimacy - Engagement in Affectionate Behaviors
Description: Measured by the Physical Intimacy Behavior scale which asks participants the frequency that they engage in affectionate behaviors answering four questions on a scale from 1 (none of the time) to 4 (most or all of the time). Scores range from 4 to 16 with higher scores indicating higher physical intimacy.
Time Frame: Baseline, 3, 6, and 12-months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 161 | 167 | 152
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 81 | 83 | 76
  Survivor: Baseline-6mo | 0.37 [-0.18 to 0.92] | 0.08 [-0.45 to 0.60] | 0.19 [-0.41 to 0.79]
  Survivor: 6mo-12mo: number analyzed (Participants) | 81 | 83 | 76
  Survivor: 6mo-12mo | -0.04 [-0.57 to 0.49] | 0.02 [-0.50 to 0.54] | 0.15 [-0.45 to 0.74]
  Partner: Baseline-6mo: number analyzed (Participants) | 80 | 84 | 76
  Partner: Baseline-6mo | 0.30 [-0.22 to 0.82] | 0.29 [-0.22 to 0.79] | 0.23 [-0.36 to 0.82]
  Partner: 6mo-12mo: number analyzed (Participants) | 80 | 84 | 76
  Partner: 6mo-12mo | -0.37 [-0.93 to 0.18] | -0.18 [-0.72 to 0.36] | -0.15 [-0.79 to 0.50]

6. Primary Outcome: Concealment of Symptoms
Description: Measured by the Emotional-Intimacy Disruptive Behavior Scale. Patients report the extent to which they engage in 8 behaviors using a scale from 1 (rarely or none of the time) to 4 (most or all of the time). Scores range from 8-32 where higher scores indicate more concealment Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -.24 [-.88 to .40] | .07 [-.56 to .69] | -.82 [-1.52 to -.11]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -.23 [-.82 to .36] | -.18 [-.77 to .41] | .53 [-.14 to 1.20]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -.33 [-.98 to .33] | -.44 [-1.07 to .22] | -.70 [-1.41 to .01]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | .63 [.04 to 1.23] | -.23 [-.82 to .36] | -.11 [-.76 to .55]

7. Primary Outcome: Pain Incongruence - Pain Intensity
Description: Measured by the degree of agreement (change or difference) between the survivor and partner ratings of the survivor's pain using the Brief Pain Inventory (BPI). This instrument has 2 subscales, pain intensity and pain interference. Values from items within each subscale are averaged together to yield scores 0-10. Low values indicate "no pain" and high values represent "pain as bad as you can imagine".
  Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Baseline-6mo | .17 [-.13 to .47] | .08 [-.22 to .37] | .16 [-.16 to .48]
  6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  6mo-12mo | -.08 [-.38 to .21] | .16 [-.14 to .44] | .16 [-.16 to .48]

8. Primary Outcome: Pain Incongruence - Pain Interference
Description: Measured by the degree of agreement (difference) between the survivor and partner ratings of the survivor's pain using the Brief Pain Inventory (BPI). This instrument has 2 subscales, pain intensity and pain interference. Values from items within each subscale are averaged together to yield scores 0-10. Low values indicate "no pain" and high values represent "pain as bad as you can imagine".
  Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Baseline-6mo | -.38 [-.70 to -.07] | .01 [-.30 to .32] | -.05 [-.38 to .29]
  6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  6mo-12mo | .27 [-.04 to .58] | -.09 [-.39 to .21] | .16 [-.17 to .50]

9. Primary Outcome: Fatigue Incongruence
Description: Measured by the degree of agreement (difference) between the survivor and partner ratings of the survivor's fatigue in the past 7 days using the Functional Assessment in Chronic Illness Therapy (FACIT) fatigue questionnaire. This instrument has 13 items, and possible scores from 0 to 52. Low values indicate no fatigue, while high values indicate high fatigue.
  Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Baseline-6mo | 1.02 [-.28 to 2.32] | -1.24 [-2.50 to .03] | -.41 [-1.80 to .98]
  6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  6mo-12mo | -1.20 [-2.49 to .10] | -.03 [-1.30 to 1.24] | -.67 [-2.08 to .74]

10. Primary Outcome: Perceived Physical Function Incongruence
Description: Measured by the degree of agreement (difference) between the survivor and partner ratings of the survivor's physical function in the past 4 weeks using the perceived physical function subscale of the SF-36 medical outcomes survey. Possible scores range from 0-100. Low scores indicate a high degree of limitation in performing physical activities, whereas high scores represent no limitations in performing physical activities due to health.
  Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Baseline-6mo | .41 [-.87 to 1.68] | -.66 [-1.90 to .59] | -.83 [-2.19 to .53]
  6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  6mo-12mo | 1.33 [.05 to 2.61] | .62 [-.64 to 1.88] | 1.29 [-.10 to 2.69]

11. Secondary Outcome: Body Composition - Bone-free Lean Mass
Description: Measured by bone-free lean (kg) for the whole body determined from a whole body dual energy x-ray absorptiometry (DXA) (Hologic-QDR Discovery Wi; APEX software, v.4.02) scan.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: kg per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
kg per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | 3.38 [2.88 to 3.88] | 3.19 [2.71 to 3.67] | 3.19 [2.61 to 3.77]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.89 [-1.38 to -0.39] | -0.60 [-1.06 to -0.14] | -1.04 [-1.59 to -0.49]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | 3.20 [2.73 to 3.67] | 3.32 [2.86 to 3.79] | 3.17 [2.62 to 3.72]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -1.43 [-1.96 to -0.90] | -1.03 [-1.53 to -0.52] | -1.05 [-1.64 to -0.46]

12. Secondary Outcome: Body Composition - Fat Mass
Description: Measured by fat mas (kg) for the whole body determined from a whole body dual x-ray absorptiometry (DXA) (Hologic-QDR Discovery Wi; APEX software, v.4.02) scan.
Time Frame: Baseline, 3, 6, and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: kg per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
kg per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -3.32 [-3.94 to -2.71] | -3.50 [-4.10 to -2.91] | -2.77 [-3.49 to -2.05]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | 1.38 [0.80 to 1.96] | 1.05 [0.52 to 1.59] | 0.53 [-0.12 to 1.18]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -3.63 [-4.17 to -3.09] | -3.36 [-3.90 to -2.83] | -3.16 [-3.79 to -2.52]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | 0.22 [-0.56 to 0.99] | 0.87 [0.14 to 1.60] | 0.25 [-0.62 to 1.11]

13. Secondary Outcome: Cardiovascular Health: Serum Cholesterol
Description: Measured by serum fasting total cholesterol.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: mg/dL per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
mg/dL per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -4.23 [-10.56 to 2.09] | 2.74 [-3.34 to 8.81] | -6.45 [-13.77 to 0.88]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | 3.77 [-3.36 to 10.89] | -0.71 [-7.11 to 5.70] | 2.68 [-4.88 to 10.24]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -2.89 [-9.71 to 3.92] | -2.18 [-11.10 to 2.74] | -2.91 [-10.70 to 4.87]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -1.30 [-8.40 to 5.79] | -3.11 [-9.94 to 3.72] | 0.85 [-6.86 to 8.56]

14. Secondary Outcome: Cardiovascular Health: Serum Triglycerides
Description: Measured by serum triglycerides.
Time Frame: Baseline, 3, 6, and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: mg/dL per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
mg/dL per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -9.86 [-22.47 to 2.65] | 7.00 [-5.01 to 19.00] | -9.76 [-23.99 to 4.46]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | 4.79 [-10.48 to 20.06] | -0.15 [-13.74 to 13.44] | 12.02 [-3.97 to 28.00]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -4.53 [-17.30 to 8.24] | 11.13 [-1.83 to 24.09] | 2.64 [-11.92 to 17.21]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -8.44 [-23.29 to 6.42] | -15.28 [-29.55 to -1.01] | 16.41 [0.29 to 32.53]

15. Secondary Outcome: Cardiovascular Health: Insulin Resistance
Description: Measured by Homeostasis Model Assessment - Insulin Resistance (HOMA-IR) - used to assess insulin sensitivity and predict the risk of type 2 diabetes and other metabolic disorders. Calculated as the product of glucose and insulin, obtained from a fasting blood sample, divided by a constant, 405. Scores generally range from 0.5 to 2.5, with lower scores indicating better insulin sensitivity and higher scores suggesting higher insulin resistance. A HOMA-IR score of 1.0 or less is considered optimal, while scores above 2.9 may indicate significant insulin resistance. Reported values reflect the estimated slope over 6-months. (Glucose mg/dL * insulin uIU/ml) / 405
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -0.06 [-0.17 to 0.06] | -0.02 [-0.13 to 0.09] | -0.01 [-0.14 to 0.12]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.05 [-0.19 to 0.01] | 0.01 [-0.13 to 0.14] | -0.03 [-0.19 to 0.12]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | 0.01 [-0.10 to 0.12] | -0.13 [-0.24 to -0.02] | 0.03 [-0.10 to 0.16]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -0.01 [-0.15 to 0.13] | 0.13 [0.00 to 0.26] | -0.08 [-0.24 to 0.07]

16. Secondary Outcome: Cardiovascular Health: Resting Systolic Blood Pressure
Description: Measured by the average of three consecutive resting blood pressure measurements (systolic and diastolic pressures).
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: mmHg per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
mmHg per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -4.91 [-7.81 to -2.00] | -5.50 [-8.31 to -2.69] | -3.34 [-6.67 to 0.00]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | 0.83 [-2.46 to 4.12] | 3.46 [0.41 to 6.51] | 2.38 [-1.25 to 6.02]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -5.92 [-9.16 to -2.67] | -7.58 [-10.8 to -4.34] | -7.93 [-11.67 to -4.19]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -0.41 [-3.58 to 2.76] | -7.02 [-12.37 to -1.67] | -1.56 [-5.14 to 2.03]

17. Secondary Outcome: Cardiovascular Health: Resting Diastolic Blood Pressure
Description: Measured by the average of three consecutive resting blood pressure measurements (systolic and diastolic pressures).
Time Frame: Baseline, 3, 6, 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: mmHg per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
mmHg per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -2.07 [-3.84 to -0.29] | -4.10 [-5.81 to -2.38] | -2.34 [-4.40 to -0.29]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | 1.42 [-0.83 to 3.67] | 1.14 [-0.95 to 3.22] | 1.48 [-1.01 to 3.97]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -3.26 [-5.29 to -1.23] | -4.93 [-6.96 to -2.90] | -2.50 [-4.87 to -0.13]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -0.58 [-2.65 to 1.49] | -1.30 [-3.31 to 0.72] | -2.26 [-4.60 to 0.09]

18. Secondary Outcome: Inflammation-hsCRP
Description: Measured by serum levels of high sensitivity C-reactive protein (hsCRP) obtained from a fasting blood sample.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: mg/L per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
mg/L per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -0.11 [-0.34 to 0.13] | 0.09 [-0.32 to 0.14] | -0.05 [-0.22 to 0.31]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.12 [-0.36 to 0.12] | -0.20 [-0.43 to 0.02] | 0.13 [-0.39 to 0.13]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | 0.01 [-0.34 to 0.13] | -0.11 [-0.32 to 0.10] | -0.04 [-0.29 to 0.22]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | -0.12 [-0.40 to 0.17] | -0.13 [-0.40 to 0.15] | -0.03 [-0.34 to 0.29]

19. Secondary Outcome: Inflammation-TNF Alpha
Description: Measured by serum levels of tumor necrosis factor alpha (TNF alpha) obtained from a fasting blood sample.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: pg/mL per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
pg/mL per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -0.01 [-0.05 to 0.03] | -0.02 [-0.05 to 0.02] | -0.03 [-0.08 to 0.01]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.01 [-0.06 to 0.04] | -0.02 [-0.07 to 0.03] | -0.01 [-0.06 to 0.05]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -0.02 [-0.06 to 0.02] | -0.02 [-0.06 to 0.02] | 0.00 [-0.05 to 0.05]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | 0.00 [-0.05 to 0.06] | 0.00 [-0.05 to 0.06] | 0.03 [-0.30 to 0.10]

20. Secondary Outcome: Objective Physical Function
Description: Measured by the Physical Performance Battery (PPB) to determine a person's ability to perform daily tasks independently. The PPB consists of 3 timed tests: 5 repeated chair stands, standing balance, and gait speed over 4 meters. Each test is scored 0 (unable) to 4 (completes without difficulty), based on quartiles of performance, then scores are summed. The possible range of scores is 0-12.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | 0.75 [0.46 to 1.04] | 0.86 [0.60 to 1.17] | 0.73 [0.41 to 1.06]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.03 [-0.27 to 0.22] | -0.07 [-0.30 to 0.15] | -0.30 [-0.57 to -0.03]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | 0.15 [-0.14 to 0.43] | 0.82 [0.54 to 1.11] | 0.73 [0.41 to 1.06]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | 0.11 [-0.13 to 0.34] | -0.18 [-0.41 to 0.05] | -0.11 [-0.38 to 0.16]

21. Secondary Outcome: Quality of Life (QOL): QLQ-C30 - Physical Functioning
Description: Measures QOL in cancer patients including subscales of physical functioning. Scores range from 0-100 for overall QOL and subscales where higher scores indicate better functioning.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are survivors only since this scale is cancer survivor specific.
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 82 | 85 | 81
Score on a scale per 6 months
  Survivor: Baseline-6mo | 2.12 [0.13 to 4.11] | 1.23 [-0.70 to 3.17] | 1.26 [-0.85 to 3.37]
  Survivor: 6mo-12mo | -1.44 [-3.56 to 0.68] | -0.30 [-2.40 to 1.80] | 1.74 [-0.63 to 4.10]

22. Secondary Outcome: Quality of Life (QOL): QLQ-C30 - Emotional Functioning
Description: Measures QOL in cancer patients including subscales of emotional functioning. Scores range from 0-100 for overall QOL and subscales where higher scores indicate better functioning.
Time Frame: Baseline, 3, 6, 12 months
Population: Overall number of participants analyzed are survivors only since this scale is cancer survivor specific.
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 82 | 85 | 81
Score on a scale per 6 months
  Survivor: Baseline-6mo | 4.18 [0.94 to 7.42] | 1.82 [-1.36 to 4.98] | 4.67 [1.26 to 8.09]
  Survivor: 6mo-12mo | -0.34 [-2.22 to 2.64] | -0.39 [-3.33 to 2.56] | -1.99 [-5.30 to 1.31]

23. Secondary Outcome: Quality of Life (QOL): SF-36 Physical Function Subscale
Description: The SF-36 measures quality of life using 8 subscales: perceived physical function, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perceptions. All subscales have possible scores from 0-100, with items from each subscale averaged together. Low scores indicate worse physical functioning, while higher scores indicate better physical functioning.
Time Frame: Baseline, 3, 6 and 12 months
Population: This measure had a significant amount of missing data for partners (due to a survey logic error) so the total sample size is reduced.
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 132 | 135 | 124
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | 1.73 [0.55 to 2.91] | 2.47 [1.33 to 3.62] | 0.96 [-0.28 to 2.20]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.76 [-1.86 to 0.34] | -0.56 [-1.65 to 0.54] | -0.81 [-2.03 to 0.40]
  Partner: Baseline-6mo: number analyzed (Participants) | 50 | 50 | 43
  Partner: Baseline-6mo | 1.81 [0.01 to 3.61] | 1.94 [0.13 to 3.76] | 0.12 [-1.83 to 2.07]
  Partner: 6mo-12mo: number analyzed (Participants) | 50 | 50 | 43
  Partner: 6mo-12mo | -0.89 [-2.24 to 0.46] | -0.04 [-1.41 to 1.33] | 1.02 [-0.47 to 2.52]

24. Secondary Outcome: Depressive Symptoms: CES-D
Description: Measured by the Center for Epidemiological Studies-Depression (CES-D) scale to determine the degree of depressive symptoms. Scores range from 0-60, with higher scores indicating more symptoms that occur at higher frequencies.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
Score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -1.50 [-2.96 to -0.04] | -0.72 [-2.14 to 0.70] | -1.10 [-2.63 to 0.44]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.10 [-1.35 to 1.16] | 0.26 [-0.99 to 1.50] | -0.21 [-1.59 to 1.18]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -1.41 [-2.65 to -0.16] | -1.73 [-2.95 to -0.52] | -1.76 [-3.11 to -0.41]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | 1.07 [-0.30 to 2.45] | -0.29 [-1.64 to 1.05] | 0.83 [-0.68 to 2.34]

25. Secondary Outcome: Anxiety: PROMIS Anxiety Short Form
Description: Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) anxiety short form 8a, using T score, standardized to mean = 50, SD = 10. Possible range for this short form is 37.1-83.1. Higher T scores reflect higher anxiety. Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are total number of individuals (survivors + partners)
Measure: Mean (95% Confidence Interval); unit: T score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 164 | 170 | 162
T score on a scale per 6 months
  Survivor: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: Baseline-6mo | -1.93 [-3.36 to -0.51] | -2.23 [-3.62 to -0.84] | -1.18 [-2.69 to 0.33]
  Survivor: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Survivor: 6mo-12mo | -0.30 [-1.80 to 1.21] | 0.42 [-1.08 to 1.91] | -0.23 [-1.89 to 1.44]
  Partner: Baseline-6mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: Baseline-6mo | -1.71 [-3.09 to -0.33] | -0.94 [-2.28 to 0.41] | -1.40 [-2.89 to 0.10]
  Partner: 6mo-12mo: number analyzed (Participants) | 82 | 85 | 81
  Partner: 6mo-12mo | 1.17 [-0.46 to 2.80] | -0.16 [-1.74 to 1.42] | -1.25 [-3.02 to 0.52]

26. Secondary Outcome: Fear of Recurrence
Description: Measured by the Fear of Recurrence scale to assess the amount of concern survivors have about their cancer returning in the future. Participants respond to 22 questions ranging from 1 (strongly agree) to 5 (strongly disagree). The possible range is 22-110. Higher scores reflect higher fear. Reported values reflect the estimated slope over 6-months.
Time Frame: Baseline, 3, 6 and 12 months
Population: Overall number of participants analyzed are survivors only since this scale is cancer survivor specific.
Measure: Mean (95% Confidence Interval); unit: Score on a scale per 6 months
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
Number analyzed (Participants) | 82 | 85 | 81
Score on a scale per 6 months
  Survivor: Baseline-6mo | -2.61 [-5.01 to -0.20] | -2.48 [-4.82 to -0.14] | -3.72 [-6.31 to -1.13]
  Survivor: 6mo-12mo | -1.63 [-3.99 to 0.73] | -1.72 [-4.04 to 0.59] | -0.31 [-2.89 to 2.28]

ADVERSE EVENTS:
Time Frame: An Adverse Event survey was created by the study team to be administered monthly during the participants' year-long participation in the study.
Arm/Group | Arm I (Supervised Exercise Together) | Arm II (Supervised Exercise Separately) | Arm III (Unsupervised Exercise Separately)
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/170 | 0/162
Serious Adverse Events (participants affected / at risk) | 4/164 | 2/170 | 1/162
Other Adverse Events (participants affected / at risk) | 9/164 | 6/170 | 3/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Supervised Exercise Together) (N=164) | Arm II (Supervised Exercise Separately) (N=170) | Arm III (Unsupervised Exercise Separately) (N=162)
Abscess - survivors (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Surgery - survivors (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1)
TIA - survivors (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Surgery - partners (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Supervised Exercise Together) (N=164) | Arm II (Supervised Exercise Separately) (N=170) | Arm III (Unsupervised Exercise Separately) (N=162)
Joint or muscle pain - survivors (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
This clinical trial enrolled couples (cancer survivors + intimate care partners), thus the information related to participant flow in the trial is reported at the couple level. Outcomes are reported at the level of the individual, thus outcome data are presented for each cancer survivors and care partners over the intervention period (baseline-6 months) and the follow-up period (6 - 12 months).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT03630354/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/54/NCT03630354/ICF_000.pdf